CLINICAL TRIAL: NCT07254494
Title: Comparative Evaluation of Resorbable (Pericardium) Versus Non Resorbable (Polytetrafluoroethylene) Membrane for Horizontal Bone Augmentation of Posterior Atrophic Mandible
Brief Title: Guided Bone Regeneration in Lower Posterior Edentulous Arch Using Resorbable or Non Resorbable Membrane.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beirut Arab University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-H-0161-D-M-0692
Record Dates: First submitted 2025-09-11; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-06

CONDITIONS: Horizontal Alveolar Bone Defect; Guided Bone Regeneration
Keywords: atrophic; horizontal bone loss; guided bone regeneration; pericardium membrane; PTFE membrane; resorbable membrane; non resorbable membrane; GBR
MeSH Terms: conditions — Atrophy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: oral pathologist
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- guided bone regeneration using Resorbable membrane pericardium (Experimental): A resorbable pericardium membrane will be fixed with titanium pins on the lingual bone plate (2-3mm from the bone crest) and on the buccal bone plate allowing for packing of particulate mix of bone graft (50% Xenograft: 50% Autogenous graft). Overfilling of the graft will be respected to compensate for future resorption. The membrane will be stretched over the graft ensuring maximum immobilization of the graft.
  Interventions: Procedure: guided bone regeneration using Resorbable membrane pericardium
- guided bone regeneration using non resorbable membrane polytetrafluoroethylene PTFE (Experimental): A non-resorbable polytetrafluoroethylene (PTFE) membrane will be fixed with titanium tacks on the lingual bone plate (2-3mm from the bone crest) and on the buccal bone plate allowing for packing of particulate mix of bone graft (50% Xenograft: 50% Autogenous graft). Overfilling of the graft will be respected to compensate for future resorption.
  Interventions: Procedure: guided bone regeneration using non resorbable ptfe membrane

INTERVENTIONS:
Procedure: guided bone regeneration using Resorbable membrane pericardium — A resorbable pericardium membrane will be fixed with titanium pins on the lingual bone plate (2-3mm from the bone crest) and on the buccal bone plate allowing for packing of particulate mix of bone graft (50% Xenograft: 50% Autogenous graft). Overfilling of the graft will be respected to compensate for future resorption. The membrane will be stretched over the graft ensuring maximum immobilization of the graft.
  Arms: guided bone regeneration using Resorbable membrane pericardium
Procedure: guided bone regeneration using non resorbable ptfe membrane — A non-resorbable polytetrafluoroethylene (PTFE) membrane will be fixed with titanium tacks on the lingual bone plate (2-3mm from the bone crest) and on the buccal bone plate allowing for packing of particulate mix of bone graft (50% Xenograft: 50% Autogenous graft). Overfilling of the graft will be respected to compensate for future resorption.
  Arms: guided bone regeneration using non resorbable membrane polytetrafluoroethylene PTFE

SUMMARY:
the purpose of this study is to compare the efficiency of non-resorbable membrane versus resorbable membrane in guided bone regeneration in atrophic posterior mandible.

DETAILED DESCRIPTION:
Lack of adequate bone for implant placement due to a previous history of periodontal disease, traumatic tooth extraction, or bone loss from prolonged use of a removable prothesis, is a common challenge in implant dentistry . Bone loss after tooth extraction has been reported to range between 40% and 60% during the first 3 years, and thereafter it is estimated to range between 0.25% and 0.5% annually .

Alveolar atrophy refers to the pathological condition where there is moderate to severe resorption of alveolar bone due to tooth loss . When teeth are lost, the functional stimulus for the alveolar bone is also lost, leading to predictable bone resorption The pattern of resorption varies based on location, where in the mandible, alveolar bone resorption is primarily horizontal, while in the interforaminal regions, it tends to be centripetal and in retroforaminal areas, the resorption is vertical and centrifugal. The presence of the inferior alveolar nerve (IAN) further complicates treatment in the posterior regions of the mandible when using Osseo integrated implants. These challenges necessitate careful planning and consideration during implant placement to achieve successful outcomes.

Various methods are employed to regenerate bone in areas with deficiencies, including using autogenous or allogeneic block grafts (cortical, cancellous, or cortico-cancellous), ridge splitting techniques, distraction osteogenesis, orthodontic tooth movement, and guided bone regeneration (GBR) with or without additional filler materials.

Numerous materials have been utilized for bone regeneration, with ongoing research in this field to address bone defects. Particularly in the context of widespread implant usage, various options such as autogenous bone, allogeneic bone, and synthetic bone have been employed to treat oral and maxillofacial bone defects . Although fresh autogenous bone yields optimal regeneration results due to its osteoinductive and osteoconductive properties, it comes with drawbacks like pain and edema from donor site injury, limited harvest volume, and high graft resorption rates. Consequently, allogeneic bone graft materials, lacking inherent bone regenerative capacity but obviating the need for an additional donor site, have gained significant use. However, due to their source from other individuals, these tissues may provoke an immune response in recipient tissues, posing a potential antigenic challenge.

Barrier membranes play a crucial role in guided bone regeneration (GBR), with various types being utilized resorbable (pericardium collagen …) and non-resorbable membrane. (e-PTFE,d-PTFE….).

Polytetrafluoroethylene (PTFE) serves as the foundational material for the most prominent and earliest non-absorbable membranes used clinically. This substance is derived from an unbranched, linear, semi-crystalline polymer comprising a combination of fluorine and carbon. PTFE falls under the category of polyhaloolefins and is classified as a thermoplastic material. Additionally, it is widely regarded for its high inertness. Titanium-reinforced membranes have been created to overcome this deficiency. A titanium skeleton with high strength and stiffness is inserted into the PTFE membrane to give it excellent plasticity and volume stability.

Several types of PTFE membrane have been introduced (e-PTFE and D-PTTFE). The e-PTFE membrane promotes tissue cell attachment and stabilizes wounds by having small pores that limit the migration of connective tissue and epithelial cells . However, its exposure to the oral cavity increases the risk of bacterial penetration and often requires premature removal, which can negatively impact outcomes . Resorbable membranes have a higher rate of resorption after exposure, leading to potential adverse effects. The ability of the e-PTFE membrane to attach to tissue often necessitates a second surgery for removal. Consequently, non-resorbable membranes are now widely used instead of e-PTFE membranes . The use of d-PTFE in dentistry is gaining acceptance due to its smaller pore size, reducing the risk of bacterial contamination when left exposed in the oral cavity. d-PTFE membranes effectively maintain space, stabilize wounds, and allow sufficient time for bone regeneration. Their non-attachment to tissue enables removal through the mucosal flap without causing trauma. Nevertheless, due to limited porosity, adequate blood supply to the area relies on marrow space and cortical perforations for successful bone regeneration

At present, titanium-reinforced membranes have become a well-established foundational material for creating stable volumes conducive to osteogenic space, thereby facilitating bone tissue regeneration in clinical settings . According to a recent meta-analysis, titanium-reinforced d-PTFE emerged as the optimal choice for guided bone regeneration (GBR) or guided tissue regeneration (GTR), as it demonstrated the highest vertical bone regeneration potential coupled with a low incidence of complications Hence, absorbable membranes that can mimic the effects of nonabsorbable ones have gained recent attention. For instance, we opted for pericardium, an absorbable membrane derived from human pericardial tissue The pericardium is a sac made of fibrous and serous tissues that envelops the heart in mammals. It has been extensively utilized in cardiac surgery for tasks such as reconstruction, repairing valves, and closing the pericardial layer. Pericardial tissue is renowned for its excellent handling properties and consistent ability to retain sutures . Furthermore, it possesses innate qualities that make it resistant to thrombosis and infection. Xenogeneic pericardium, sourced mainly from bovine and porcine origins, and occasionally from equine sources, is commonly used. These tissues are available in large patches, allowing for customized shaping to suit various cardiovascular procedures. Predominantly composed of collagen fibers, xenogeneic pericardium possesses elastic properties, enabling it to adapt to intricate anatomical structures.

The selection of an appropriate tissue barrier involves considering various properties of the pericardium membrane. These include its physical characteristics, biocompatibility, biodegradability, immunogenicity, capacity to attract and stimulate periodontal ligament fibroblast cells, as well as its ability to promote adherence and proliferation of regenerative cells. Additionally, the membrane's potential to effectively seal the underlying defect is crucial for its success. Pericardium membranes have demonstrated strong crosslinking, suggesting a longer duration for resorption.

Additionally, the pericardium membrane provides a scaffold for attachment, migration, and proliferation of periodontal ligament fibroblasts, thereby promoting regeneration of soft tissues. As part of guided bone regeneration, the pericardium membrane facilitates the release of growth factors and preserves blood supply to the affected area, thereby promoting growth of bone and soft tissue and enabling regeneration of periodontal tissues.

Pericardium has found widespread use in regenerating bone defects around implants or serving as a barrier membrane for maxillary sinus perforations. However, there remains a scarcity of clinical studies assessing these procedures.

In this context, the purpose of this study is to compare the efficiency of non-resorbable membrane versus resorbable membrane in guided bone regeneration in atrophic posterior mandible.

Null hypothesis is that there is no significant difference between the pericardium and the d-PTFE membrane.

The primary objective of this study is to evaluate and compare clinically, radiographically, and histologically the efficiency of native pericardium porcine collagen membrane (Botiss Jason®) versus d-PTFE non resorbable membrane for horizontal augmentation of alveolar ridge for patients with posterior mandibular atrophy. Twenty partially edentulous patients with horizontal bone deficiency in the posterior mandibular ridge requiring bone augmentation and implant-supported restoration who will be referred to the Periodontal department in the faculty of dentistry at Beirut Arab university, Lebanon, will be included in the protocol. Subjects will be randomly assigned to one of 2 groups: controls (group A:10) who will receive GBRB using d-PTFE barrier, and experimental (group B:10) who will receive GBR using native pericardium collagen membrane. Subjects from both groups will be treated with the selected barrier and the underlying space-making composite graft of xenograft plus autogenous bone to help support the overlying membrane.

Inclusion criteria:

1. Both males and females of age 18 years or older
2. Mandibular posterior atrophic alveolar ridge Required horizontal bone augmentation procedures prior to implant placement.
3. Alveolar bone height suitable for implant placement.
4. Free of any local or systemic condition that may contraindicate ridge expansion procedure
5. The capacity to understand and accept the conditions of the study.
6. Continuing participation over at least 1 year of follow-up. Exclusion criteria

1. Heavy smokers (i.e., 2 or more packs of cigarettes per day); 2. Insufficient oral hygiene 3. Acute local or systemic infection 4. Patients with any systemic disease that may affect bone healing; 5. Pregnancy or the possibility of becoming pregnant during the study; and 6. Addiction to drugs or alcohol Methods

All the patients will be subjected to the pre surgical phase which include:

1. Patient history:

   1. Personal history
   2. Past medical and dental history
2. Clinical and radiographic examination

   1. Both extra and intra oral examination will be done
   2. A routine panoramic x-ray for patient selection
   3. A CBCT x-ray for preoperative implant site assessment
3. Phase 1 therapy:

   a. Plaque control education: i. Diet control (in patient with rampant caries) ii. Removal of calculus and root planning iii. Correction of restorative and prosthetic irritation factors iv. Excavation of caries and restoration (temporary or final, depending on whether a definitive prognosis for the tooth has been determined and location of caries) v. Antimicrobial therapy (local or systemic if needed) b. Each patient will undergo oral hygiene measures such as electronic scaling, polishing and mouthwash usage for a couple days.
4. Surgical phase

   1. Patient preparation:

      * Extraoral scrubbing with 5% povidone-iodine solution.
      * The patient's mouth will be rinsed with a solution of chlorhexidine digluconate 0.2% for 2 minutes.
   2. Surgical procedures STAGE 1

      * A local anesthetic will be administered using 4%lidocaine hydrochloride.
      * A mid-crestal horizontal incision within the keratinized tissue of the edentulous ridge.
      * A vertical incision will be made to coronally advance the flap.
      * A periosteal release of the flap will be performed.
      * A dissection will be made to remove the tension and muscle fibers in the flap in order to have a tension free and a coronally advanced flap.
      * Cortical perforations will be made with #8 round bur.
      * 8-mm tenting screws will be placed with 3 mm incorporated into the bone.
      * Bone harvesting using a bone scraper.
      * Creation of 50:50 bone mixtures of xenograft and autogenous bone placement
      * Lingual fixation of ti-reinforced d-PTFE membranes (cytoplast ti-250xl; osteogenics biomedical) in group A or fixation of pericardium native collagen membrane (jason membrane) in group B.
      * Filling and adaptation of the biomaterial mixture under the membrane.
      * Buccal-side fixation using two or three mini-screws (pro-fix membrane fixation screws)
      * Free-tension primary closure using double-line suturing by PTFE (4-0) sutures, and PGA sutures (4-0 and 6-0)
      * Written postoperative instructions and medications will be given to the patients. These include amoxicillin 500 mg tablets, hydrocodone/APAP 10/325, 0.12% chlorhexidine solution, and ibuprofen 600 mg, chlorhexidine gluconate mouth rinse (0.12% t.i.d.), and topical chlorhexidine 4 times per day applied to the surgical site.

Cone Beam Volumetric Topography (CBVT). Two CBVT, one before and one after 6 months will be recorded with the previously used acrylic template with a radiopaque indicator in place. One single examiner who will be blinded and calibrated for the procedures will evaluate the images. For the calibration, the examiner will evaluate 10 images 2 times within 24 hours apart and will measure the primary outcome, i.e. horizontal bone thickness. The agreement of the measurements will be assessed with the intra-class correlation. The following measures will be assessed: 1) Horizontal bone thickness, measured in 3 levels (3, 5, and 7mm distant from the bone crest); 2) Bone Height, the distance between the bone crest and a fixed reference point; 3) Horizontal and Height Bone Gain, the variation between baseline and the final measures of both parameters (Δ=final-initial). In addition, the volume of bone gain will be assessed.

Patient-centred outcomes. Postoperative pain and discomfort and analgesic consumption will be assessed using a questionnaire during the following 7 postoperative days. The patients will be requested to monitor their postoperative pain/discomfort and the number of days on analgesics during this period.

Histological analysis. After 6 months, the site will be re-opened. The flap outline will be similar to the first surgery. The surgical access will be limited to the crestal area except for group 3. Titanium screws will be removed in group 1. Non-resorbable membrane and pseudo-membrane layer will be removed in group 3. A 2mm trephine bur will be used to collect a core biopsy at the preplanned implant positions for histomorphometric analysis. Root-form dental implants will be placed with the proper lengths and diameters. Area and percentage of areas will be assessed for the newly formed bone, the bone marrow spaces, and bone graft particles.

Clinical measurement: the frequency of complications, i.e. episodes of suppuration, membrane exposure, and suture dehiscence, will be recorded. In addition, the implant insertion torque will be evaluated.

Statistical analyses Descriptive statistics will be expressed as mean ± standard deviation and percentage. Normality will be tested using the Shapiro-Wilk test. Values referring to VAS scores will be compared using One-way ANOVA (Wilcoxon in case of the non-normal distribution data), the horizontal bone gain will be assessed with Repeated Measures of Variance. The frequency of sites effects will be assessed with X2. For the histological analyses, the volume of vital bone, graft remnants, and connective tissue will be measured based on the averages of the percentages and compared using One-way ANOVA (Wilcoxon in case of the non-normal distribution data). A significance of 5% will be used for all analyses.

ELIGIBILITY:
Inclusion Criteria:

* Mandibular posterior atrophic alveolar ridge Required horizontal bone augmentation procedures prior to implant placement.
* Alveolar bone height suitable for implant placement.
* Free of any local or systemic condition that may contraindicate ridge expansion procedure
* The capacity to understand and accept the conditions of the study.
* Continuing participation over at least 1 year of follow-up.

Exclusion Criteria:

* Heavy smokers (i.e., 2 or more packs of cigarettes per day);
* Insufficient oral hygiene
* Acute local or systemic infection
* Patients with any systemic disease that may affect bone healing;
* Pregnancy or the possibility of becoming pregnant during the study; and
* Addiction to drugs or alcohol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Osstell Implant Stability Quotient (ISQ) | 6 months after the surgery at the time of implant placement
  measure the implant stability in both group using osstell machine ,The ISQ scale ranges from 1 to 99, with higher values indicating greater stability
change from baseline in pain as measured by the visual analogue scale VAS | baseline,12 weeks
  pain sensation measured by VAS visual analogue scale score of both group the VAS ranges from 0 to 100 with 0 indicating no pain and higher scores indicating greater pain. scores are measured on a 100 mm VAS

SECONDARY OUTCOMES:
Horizontal bone gain measured using CBCT in mm | 6 months
  Participants will undergo radiographic evaluation using cone-beam computed tomography (CBCT) performed preoperatively, immediately post-operatively, and six months post-operatively. Linear horizontal ridge width will be measured at standardized reference points on the CBCT scans using digital caliper measurement tools within the CBCT analysis software. The outcome will assess the amount of horizontal bone gain (in millimeters) achieved following the augmentation procedure.
Qualitative bone assessment using histological and histomorphometric analysis to measure the % of bone | 6 months
  A core biopsy will be obtained from the grafted site six months post-operatively to evaluate the quality of regenerated bone. The specimen will undergo histological and histomorphometric analysis using standard light microscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Beirut arab university, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in the publication will be made available after de-identification. Data may include [specify: e.g., demographic information, outcome measures, etc.].
Time Frame: Beginning [e.g., 6 months] after publication and continuing for [e.g., 2 years].

DOCUMENTS (1):
  • Study Protocol (2024-09-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT07254494/Prot_000.pdf